CLINICAL TRIAL: NCT06959108
Title: Randomized Phase 2 Trial of Induction Treatment of Anti-PD-1 Pucotenlimab and EGFR-ADC MRG003 Versus EGFR-ADC Alone Followed by Chemoradiotherapy in Locally Advanced Head and Neck Squamous Cell Carcinoma (LA-SCCHN).
Brief Title: Clinical Trial Comparing Induction Treatment With EGFR-ADC MRG003 Alone or in Combination With the Anti PD1 Pucotenlimab, Followed by Radiochemotherapy in Locally Advanced Squamous Cell Cancers of the Head and Neck
Acronym: IDEAL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Lepu Medical Technology (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2024-03; 2023-510558-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-04

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pucotenlimab-MRG003 (Experimental): * Induction treatment (9 weeks): 3 cycles of the anti-PD-1 Pucotenlimab in combination with the EGFR ADC MRG003
  * Concurrent chemoradiation (7 weeks). The CRT will start within 28 ± 7 days after the Day 1 of the third cycle of the EGFR ADC MRG003.
  * Adjuvant treatment (24 weeks from one month after the end of CRT).
  Interventions: Drug: Pucotenlimab; Drug: MRG003
- MRG003 alone (Active Comparator): * Induction treatment ( 9 weeks): 3 cycles of the EGFR ADC MRG003 alone
  * Concurrent chemoradiation (7 weeks). The CRT will start within 28 ± 7 days after the Day 1 of the third cycle of the EGFR ADC MRG003.
  Interventions: Drug: MRG003

INTERVENTIONS:
Drug: Pucotenlimab — 200mg every 3 weeks (21-day cycles) for a total of 3 cycles.
  Arms: Pucotenlimab-MRG003
Drug: MRG003 — 2.3 mg/kg, every 3 weeks (21-day cycles) for a total of 3 cycles.

SUMMARY:
The primary objective of this study is to compare the objective response rate (ORR) of patients with LA-HNSCC, treated with induction of EGFR-ADC MRG003 and anti PD-1 Pucotenlimab versus EGFR-ADC MRG003 alone before chemoradiotherapy.

People eligible to participate in this study must be between the ages of 18 and 75 and have locally advanced squamous cell carcinoma of the head and neck requiring treatment with chemoradiotherapy (cisplatin combined with radiotherapy).

Half of the research participants will receive MRG003 alone as induction before radiochemotherapy and the other half will receive MRG003 combined with pucotenlimab as induction before radiochemotherapy, then pucotenlimab as adjuvant* after radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Evaluable tumor burden assessed by H&N-computed tomography scan (CT-scan) or magnetic resonance imaging (MRI), based on RECIST v 1.1
* Patients eligible to cisplatin-based chemotherapy
* No hearing loss by clinical assessment or ≤ grade 2 hearing impairment (according to NCICTCAE v.5
* No prior treatment with chemotherapy, immunotherapy and targeted therapy for H&N cancer, radiotherapy or surgery in the head and neck region.

Exclusion Criteria:

* Metastatic disease (stage IVC as per AJCC/TNM, 8th Ed.).
* Patients having received prior therapy with anti-PD1, anti-PD-L1, anti-PD-L2, anti- CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting Tcell co-stimulation or checkpoint pathways).
* Treatment for other diseases with an investigational agent or use of an investigational device within 4 weeks of the first dose of study treatment
* History of another malignancy within the last 3 years prior to randomization, with the exception of completely resected non-melanoma cell skin cancer outside the head and neck area or completely resected stage I breast cancer, or completely resected in-situ nonmuscular invasive bladder, cervix, uterine and/or prostate (Gleason 6) carcinomas, or T1a squamous cell carcinoma of the esophagus or rectum/anus.
* Patients with clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication, or known persistent reduced left ventricular ejection fraction < 50%.
* Patients with positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Patients with positive tests for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection. Presence of other serious liver diseases, including chronic autoimmune hepatic disorders, primary biliary cirrhosis or sclerosing cholangitis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
objective response rate | around 20 months after the inclusion of the 1st patient
  objective response rate evaluated by the investigators with head and neck radiological imaging according to RECIST version 1.1 criteria at the end of induction phase of EGFR-ADC MRG003 + anti-PD-1 Pucotenlimab or EGFR-ADC MRG003 alone

SECONDARY OUTCOMES:
Progression-free survival | 1 year from the inclusion of the last patient
  Progression-free survival (PFS) as the time from randomization to the first progression (locoregional/metastatic progression after induction, CRT or adjuvant treatment) or death from any cause, or the date of the last follow-up for patients who did not have progression or death
Failure-free survival | 1 year from the inclusion of the last patient
  Failure-free survival (FFS) as the time from randomization to the first of the following events: locoregional /metastatic progression after the completion of CRT or failure to receive CRT; or death from any case or the date of the last follow-up for patients who did not have these events
Overall survival | 1 year from the inclusion of the last patient
  Overall survival (OS) defined as the time between randomization and death from any cause or date of the last follow-up for patients alive

CONTACTS AND LOCATIONS:
Overall Officials: Jean BOURHIS, Medical Director, Study Director — GORTEC

IPD SHARING:
Plan to Share IPD: Yes
Data collected in the eCRF
Supporting Information: Study Protocol, ICF
Time Frame: At the end of the study and the delay will be defined in the contract
Access Criteria: Researchers could be access to clinical data for participants